CLINICAL TRIAL: NCT01138787
Title: CASTELL = Cholesterol Absorption Study STErols (LL)
Brief Title: Cholesterol Absorption Inhibition Study
Acronym: CASTELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Yvonne E.M.P. Zebregs, MSc, Unilever R&D Vlaardingen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 09030V
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cholesterol Absorption Inhibition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reference spread (Active Comparator): 2250 mg PS (as PSE) in spread (30 g)
  * 50 mg labeled D7-cholesterol,
  * 30 mg 3,4-13C-cholesterol, iv dosed at same time.
  Interventions: Dietary Supplement: Reference spread
- Placebo spread (Placebo Comparator): regular light margarine (30 g)
  * 50 mg labeled D7-cholesterol,
  * 30 mg 3,4-13C-cholesterol, iv dosed at same time.
  Interventions: Dietary Supplement: Placebo spread
- Test spread (Experimental): 2250 mg PS in innovatively processed spread (30 g)
  * 50 mg labeled D7-cholesterol,
  * 30 mg 3,4-13C-cholesterol, iv dosed at same time.
  Interventions: Dietary Supplement: Test spread

INTERVENTIONS:
Dietary Supplement: Reference spread — Single dose (30 gr) of spread, containing 2250 mg PS
  Arms: Reference spread
Dietary Supplement: Placebo spread — Single dose (30 gr) of regular light margarine
  Arms: Placebo spread
Dietary Supplement: Test spread — Single dose (30 gr) of innovatively processed spread containing 2250 mg PS.
  Arms: Test spread

SUMMARY:
Rationale: Consuming Plant Sterols (PS) fortified foods is widely accepted as easy to apply, life-style change to combat modestly elevated plasma cholesterol concentrations. PS are typically formulated as PS fatty acid ester (PSE) from margarines. In this study, PS will be formulated in a new innovative type spread. To confirm that the new spread results in a comparable cholesterol absorption inhibition as the reference product a dual isotope cholesterol study is planned, prior to any larger efficacy study.

Primary objective: Cholesterol absorption inhibition (%) calculated from plasma concentration vs. time curves from labeled cholesterol, for the PS or PSE containing products, compared to a control product without PS or PSE.

Secondary objectives: PK parameters for cholesterol as derived from the plasma concentration vs. time curves.

Study design: Acute, single dose, double-blind, randomized, cross-over. Study population: 18 healthy, non-obese men (BMI 20-27 kg∙m-2, age range 20 - 65 yr) Test products: PS (2250 mg) formulated in innovatively processed spread (30 g); PSE (2250 mg PS) reference product (30 g); Control product without PS or PSE (30 g) Intervention: Three study periods during which a single dose of either Test, Reference or Control (regular light spread) spreads will be consumed together with standard breakfast. At each study period, 50 mg of D7-cholesterol is added to the meal and 30 mg of 13C-cholesterol is injected to measure cholesterol absorption. Before and four times after consumption of each spread, blood samples will be taken at 24 h intervals up to 7 days.

Key parameters: Enrichments of labeled cholesterol isotopes as determined by GCMS and IRMS. Fractional absorption is determined by the ratio of the two isotopes in plasma cholesterol after 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy: no medical conditions which might effect study measurements (judged by study physician).
2. Males aged 20 - 65
3. BMI 20-27 kg∙m-2
4. LDL-C levels between 3.0 - 5.0 mmol/L, triglycerides < 3.0 mmol/L
5. Not more than 10 hours per week of strenuous exercise
6. Ability to give informed consent.
7. Ability to follow verbal and written instructions.
8. Non-smoker (tobacco, marijuana).
9. The ability to attend and to commute to the performance site for each of study day visit and follow-up throughout the study period are required.
10. Willing to consume a breakfast in the morning of each study day.
11. Willing to consume margarine on each study occasion.
12. Having a general practitioner.
13. No use of medication which interferes with study measurements (as judged by the study physician).
14. Agreeing to be informed about medically relevant personal test-results after the screening visit by a physician.
15. Consumption =< 21 alcoholic drinks in a typical week.
16. No blood donation 1 month prior to pre-study examination or during the study.
17. Has accessible veins on the forearm as determined by examination at screening.
18. Not being an employee of Unilever.
19. No reported participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study.
20. No reported participation in night shift work during the study.

    Exclusion Criteria:
21. Unwilling to refrain from consumption of plant sterol or stanol containing products one week before and during the study..
22. Plasma lipid profile which indicates deviating lipid / cholesterol homeostasis, to be judged by study physician.
23. Evidence of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hemato¬logical/ immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/ connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/ psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol.
24. Gastrointestinal or hepatic disorders influencing gastrointestinal absorption or transit, including gallstones or biliary diseases.
25. History of surgery related to the gastro-intestinal tract
26. On a medically prescribed or weight reduction diet
27. Recreational (intravenous) drug use.
28. The use of psychotropic drugs, including: benzodiazepines or alcohol in excess of 21 units/ week for males
29. Concomitant medication that may modulate gastro-intestinal secretions and pH (e.g. antacids, proton-pump-inhibitors, prostaglandins, anticholinergic agents, H2-receptor antagonists)
30. Concomitant medication that can alter gastric emptying (e.g. metoclopramide, cisapride, domperidone and erythromycin, anticholinergics, tricyclic antidepressants, narcotic analgesics, adrenergic agents, calcium channel blockers)
31. Concomitant medication that can alter intestinal transit (e.g. loperamide, chemical/ osmotic/bulk laxatives), or influence satiety/energy intake (e.g. sibutramine, gluco¬corticoids, anabolic steroids)
32. Intolerance or allergy for test product.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
cholesterol absorption calculated from plasma cholesterol enrichments vs. time curves | 5 blood samples within one week for each intervention

SECONDARY OUTCOMES:
PK parameters derived from plasma curves (Cmax, Tmax, cholesterol pool, flux). | 5 blood samples within one week for each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maud N Vissers, Dr. Ir, Principal Investigator — Academisch Medisch Centrum, afdeling vasculaire geneeskunde; Guus SM Duchateau, Dr, Study Director — Unilever Research & Development Vlaardingen
Locations (1):
- Academisch Medisch Centrum, vasculaire geneeskunde, Amsterdam, North Holland, Netherlands